CLINICAL TRIAL: NCT06331169
Title: A Prospective Phase Ib Study of Anlotinib With Trastuzumab Deruxtecan for HER2-Low Unresectable and/or Metastatic Breast Cancer (ALTER-BC-Ib-01)
Brief Title: Anlotinib With Trastuzumab Deruxtecan for Previously Treated HER2-Low Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Director of Phase I Clinical Trial Department; Professor, Chief physician of oncology department, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-BC-Ib-01
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anlotinib dose escalation + trastuzumab deruxtecan (Experimental): Various doses of anlotinib (8 mg QD, 10 mg QD, and 12 mg QD) administered during dose escalation to determine the recommended phase 2 Dose (RP2D) + trastuzumab deruxtecan 5.4 mg/kg.
  Anlotinib at the RP2D + trastuzumab deruxtecan 5.4 mg/kg combination therapy
  Interventions: Drug: Anlotinib; Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Anlotinib — Anlotinib is a new, orally administered tyrosine kinase inhibitor that targets vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR), platelet-derived growth factor receptors (PDGFR), and c-kit.
  Other Names: Anlotinib dihydrochloride
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan is an antibody-drug conjugate composed of an anti-HER2 (human epidermal growth factor receptor 2) antibody, a cleavable tetrapeptide-based linker, and a cytotoxic topoisomerase I inhibitor.
  Other Names: DS-8201

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of anlotinib and trastuzumab deruxtecan in human epidermal growth factor receptor 2 (HER2)-low unresectable and/or metastatic breast cancer who had received ≤1 line of prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 - 75 years; ECOG PS 0 or 1. 2. Pathologically documented breast cancer that:

  1. Is unresectable or metastatic.
  2. Has a history of low HER2 expression (IHC 1+& IHC 2+/ISH- or 0<IHC<1+).
  3. Is HR-positive or HR-negative.
  4. Has progressed on, and would no longer benefit from, endocrine therapy.
  5. Has been treated with ≥1 prior lines of chemotherapy/adjuvant in the recurrent or metastatic setting.

     3. At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors version 1.1（Previously treated lesions with radiotherapy or focal therapy and no progression cannot be included as target lesion for assessment）.

     4. Has protocol-defined adequate bone marrow, renal, hepatic and blood clotting functions.

     5. Male and female subjects of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and after the last dose for at least 6 months.

     Exclusion Criteria:
     1. Has previously been treated with anti-angiogenic targeted small molecule therapy.
     2. Prior treatment with antibody drug conjugate with a topoisomerase I inhibitor exatecan derivative.
     3. Has a history of (noninfectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
     4. Has unresolved toxicities from previous anticancer therapy.
     5. Has uncontrolled or significant cardiovascular disease.
     6. Has any bleeding event, unhealed wounds, ulcerative or fractures.
     7. Has arterial or venous thromboembolic events occurred within 6 months.
     8. Has spinal cord compression or clinically active central nervous system metastases.
     9. Has any other condition that per protocol or in the opinion of the investigator is inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Determination of the RP2D of anlotinib in combination with trastuzumab deruxtecan | up to 1 year
  The RP2D is defined as the dose level for the dose expansion phase, based on safety, tolerability, efficacy collected during the dose escalation portion of the study.
Objective Response Rate (ORR) | Up to approximately 3 years
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Duration of Response (DCR) | Up to approximately 3 years
  DCR is defined as the percentage of cases with remission (PR+CR) and stable disease (SD) after treatment in the evaluable cases.
Duration of Response (DOR) | Up to approximately 3 years
  DOR is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from the participant's first dose of study treatment to the first date of either disease progression or death, whichever occurs first.
Overall Survival (OS) | Up to approximately 3 years
  OS is defined as the time from the participant's first dose of study treatment to the date of death.
Number of Participants With Adverse Events (AEs) | Up to approximately 3 years
  Assessment of the toxicity profile of regimen according to the National Cancer Institute Common Toxicity Criteria version 5.0 (NCI CTCAE v 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Jian Zhang, Shanghai, Shanghai Municipality, China